CLINICAL TRIAL: NCT07264049
Title: Education, Research, and Community Engagement Through a Food Survey [Educación, Investigación y Vinculación Con el Medio Mediante Una Encuesta Alimentaria]
Brief Title: Education and Community Engagement Through a Food Survey
Acronym: Impacta
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Finis Terrae University (Other)
Responsible Party: Principal Investigator, Layla Simon, Principal Investigator, Finis Terrae University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 24-042; Finis Creacion (Other Grant/Funding Number: FinisTerraeU)
Record Dates: First submitted 2025-11-20; First posted 2025-12-04 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Feeding Behaviors; Mental Health
Keywords: food; health; students; wellbeing; nutrition
MeSH Terms: conditions — Feeding Behavior; Psychological Well-Being | interventions — Educational Status; Nutritional Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Other): Students were educated in the relevance of feeding behaviours and nutrition in wellbeing and mental health. The book "Eat healthily" [Comer saludablemente] was written to give information of nutrition and health and to provide recepes to prepare healthy food. Cook classes and healthy breaks were aplied. Additionaly, the association between mental health and ultra procesed food consumtion was analyzed to raise awareness about this problem.
  Interventions: Other: Education in nutrition

INTERVENTIONS:
Other: Education in nutrition — Students were educated in the relevance of feeding behaviours and nutrition in wellbeing and mental health. The book "Eat healthily" [Comer saludablemente] was written to give information of nutrition and health and to provide recepes to prepare healthy food. Cook classes and healthy breaks were aplied. Additionaly, the association between mental health and ultra procesed food consumtion was analyzed to raise awareness about this problem.

SUMMARY:
The objective of this study is to conduct educational, research, and community outreach activities through the implementation of a dietary survey to improve the quality of these areas, train better professionals, and have a positive impact on people's quality of life and health.

If participants agree to participate, participants will be asked to do the following:

* Complete a dietary survey asking about the foods and beverages participants ate yesterday, and a well-being survey asking about their feelings and thoughts over the past few weeks.
* The surveys will be conducted using the DEMO ASA24® and REDCap tools. Participants will record the meals, foods, and beverages, times, quantities, and locations where participants ate the food their ate the day before from 12:00 a.m. to 11:59 p.m., as well as their feelings and thoughts over the past few weeks.
* This survey will be conducted at Finis Terrae University.
* This will take less than 30 minutes and will be completed once.
* The interviewer will access the DEMO ASA24® and REDCap platforms via a link from a mobile device or tablet connected to the university's Wi-Fi network.

DETAILED DESCRIPTION:
The objective of this study is to conduct educational, research, and community outreach activities through the implementation of a dietary survey to improve the quality of these areas, train better professionals, and have a positive impact on people's quality of life and health.

If participants agree to participate, participants will be asked to do the following:

* Complete a dietary survey asking about the foods and beverages participants ate the day before, and a well-being survey asking about their feelings and thoughts over the past few weeks.
* The surveys will be conducted using the DEMO ASA24® and REDCap tools. Participants will record the meals, foods, and beverages, times, quantities, and locations where participants ate the food participants ate the day before from 12:00 a.m. to 11:59 p.m., as well as their feelings and thoughts over the past few weeks.
* This survey will be conducted at Finis Terrae University.
* This will take less than 30 minutes and will be completed once.
* The interviewer will access the DEMO ASA24® and REDCap platforms via a link from a mobile device or tablet connected to the university's Wi-Fi network.

Participants will not benefit from participating in this research. However, the information obtained through their participation will be useful for learning more about nutritional profiles and improving the quality of life of the university community.

This research has no risks or costs to participants.

The information obtained will be kept confidential.

The results obtained may be presented in journals and conferences; however, participants name will not be disclosed.

The results obtained from this survey may be used for this study and other subsequent studies that adhere to the objective of this study.

The participation in this research is completely voluntary. The participation does not imply any benefit or adverse impact on participants academic development.

Participants have the right to decline participation or withdraw their consent and withdraw from this research at any time participants deem appropriate. By doing so, participants do not lose any rights they have as a student at this institution.

If participants withdraw their consent, participants results will be deleted and the information obtained will not be used.

Participants will be educated in the relevance of feeding behaviours and nutrition in wellbeing and mental health. The book "Eat healthy" ["Comer saludablemente"] will give information of nutrition and health and to provide recepes to prepare healthy food. Cook classes and healthy breaks will be aplied. Additionaly, the association between mental health and ultra procesed food consumtion will be analyzed to raise awareness about this problem.

ELIGIBILITY:
Inclusion Criteria:

* University students
* Time and availability to answer the reports
* Accept to participate in this study

Exclusion Criteria:

* NA

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2025-04-01 (Actual); Primary Completion 2025-04-01 (Actual); Study Completion 2025-09-28 (Actual)

PRIMARY OUTCOMES:
Nutritional profile | 3 months
  Nutritional profile through ASA24 report
Mental health | 3 months
  Mental wellbieng was analyzed through the Edinburgo test

CONTACTS AND LOCATIONS:
Locations (1):
- Finis Terrae University, Santiago, Chile

IPD SHARING:
Plan to Share IPD: No
This information is confidential